CLINICAL TRIAL: NCT01959711
Title: Randomized Clinical Trial of Posterior Retroperitoneoscopic Adrenalectomy Versus Lateral Transperitoneal Laparoscopic Adrenalectomy With a Five-year Follow-up
Brief Title: Randomized Clinical Trial of Posterior Retroperitoneoscopic Adrenalectomy Versus Lateral Laparoscopic Adrenalectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Marcin Barczynski, Associate Professor of Surgery at the Third Chair of General Surgery, Jagiellonian University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BBN 501/ZKL/130/L
Record Dates: First submitted 2013-10-06; First posted 2013-10-10 (Estimated); Last update posted 2013-10-10 (Estimated); Status verified 2013-10

CONDITIONS: Adrenal Tumor; Pheochromocytoma; Conn's Syndrome; Cushing's Syndrome
Keywords: Lateral transperitoneal laparoscopic adrenalectomy; Posterior retroperitoneoscopic adrenalectomy
MeSH Terms: conditions — Adrenal Gland Neoplasms; Pheochromocytoma; Hyperaldosteronism; Cushing Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Posterior RA (Experimental): Posterior retroperitoneoscopic adrenalectomy
  Interventions: Procedure: Posterior RA
- Lateral transperitoneal LA (Active Comparator): Lateral transperitoneal laparoscopic adrenalectomy
  Interventions: Procedure: Lateral transperitoneal LA

INTERVENTIONS:
Procedure: Posterior RA — Posterior retroperitoneoscopic adrenalectomy
  Arms: Posterior RA
Procedure: Lateral transperitoneal LA — Lateral transperitoneal laparoscopic adrenalectomy
  Arms: Lateral transperitoneal LA

SUMMARY:
Laparoscopic adrenalectomy has become the gold standard operation for non-malignant adrenal tumors replacing open adrenalectomy. The most popular lateral transperitoneal laparoscopic adrenalectomy (LTLA) approach has been recently challenged by an increasing popularity of the posterior retroperitoneoscopic adrenalectomy (PRA) approach which is believed by many surgeons as an easy to learn, reproducible and beneficial for patients. However, this belief is not evidence-based, so far. The aim of this study is to clarify if PRA is superior to the LTLA as minimally invasive approach to small and benign adrenal tumors.

DETAILED DESCRIPTION:
Laparoscopic adrenalectomy has replaced open adrenalectomy as the standard operation for non-malignant adrenal tumours. Thanks to the popularization of the posterior technique described by Walz and co-workers, the posterior retroperitoneal adrenalectomy (PRA) is being performed in increasing numbers worldwide. Advocates for the laparoscopic and retroperitoneoscopic approaches cite the advantages of each technique, but there is no published evidence that supports the superiority of one over the other. Most of the published literature is retrospective, with inadequate or no controls and with potential biases.

The aim of this study is to test the hypothesis that PRA is superior to the lateral transperitoneal laparoscopic adrenalectomy (LTLA) as minimally invasive approach to small and benign adrenal tumors.

For a sample size calculation an assumption was made that a 20% reduction in duration of surgery represents clinically relevant difference. To detect this, it was calculated that 24 patients would be required in each treatment arm to give the study a power of 90 per cent. Anticipating a 25% loss to follow-up, 32 patients per arm were required in the study.

ELIGIBILITY:
Inclusion Criteria:

* unilateral adrenal tumor below 7cm in diameter without suspicion for malignancy

Exclusion Criteria:

* active malignancy
* pregnancy or lactation
* age below 18 years, or above 80 years
* high-risk patients according to the American Society of Anesthesiology (ASA 4 grade or higher
* inability to comply with the scheduled follow-up protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2006-01; Primary Completion 2008-06 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
duration of surgery | intraoperatively

SECONDARY OUTCOMES:
postoperative recovery | participants will be followed for the duration of hospital stay, an expected average of 7 days
  including: postoperative pain, length of hospital stay, time to oral intake, time to ambulation
blood loss | participants will be followed for the duration of hospital stay, an expected average of 7 days
postoperative complications | up to 5 years after surgery
  including: pneumothorax/haemothorax, surgical emphysema, chest infection, visceral injury, peritonitis/abscess, wound infection, neuralgia, and surgical access site herniation

CONTACTS AND LOCATIONS:
Overall Officials: Marcin Barczyński, MD, PhD, Principal Investigator — Jagiellonian University
Locations (1):
- Jagiellonian University, Medical College, Third Chair of General Surgery, Krakow, Poland

REFERENCES:
- [Background] Barczynski M, Konturek A, Golkowski F, Cichon S, Huszno B, Peitgen K, Walz MK. Posterior retroperitoneoscopic adrenalectomy: a comparison between the initial experience in the invention phase and introductory phase of the new surgical technique. World J Surg. 2007 Jan;31(1):65-71. doi: 10.1007/s00268-006-0083-8. PMID 17180554
- [Background] Lee CR, Walz MK, Park S, Park JH, Jeong JS, Lee SH, Kang SW, Jeong JJ, Nam KH, Chung WY, Park CS. A comparative study of the transperitoneal and posterior retroperitoneal approaches for laparoscopic adrenalectomy for adrenal tumors. Ann Surg Oncol. 2012 Aug;19(8):2629-34. doi: 10.1245/s10434-012-2352-0. Epub 2012 Apr 20. PMID 22526902
- [Background] Perrier ND, Kennamer DL, Bao R, Jimenez C, Grubbs EG, Lee JE, Evans DB. Posterior retroperitoneoscopic adrenalectomy: preferred technique for removal of benign tumors and isolated metastases. Ann Surg. 2008 Oct;248(4):666-74. doi: 10.1097/SLA.0b013e31818a1d2a. PMID 18936580
- [Background] Walz MK, Alesina PF, Wenger FA, Deligiannis A, Szuczik E, Petersenn S, Ommer A, Groeben H, Peitgen K, Janssen OE, Philipp T, Neumann HP, Schmid KW, Mann K. Posterior retroperitoneoscopic adrenalectomy--results of 560 procedures in 520 patients. Surgery. 2006 Dec;140(6):943-8; discussion 948-50. doi: 10.1016/j.surg.2006.07.039. PMID 17188142
- [Background] Constantinides VA, Christakis I, Touska P, Palazzo FF. Systematic review and meta-analysis of retroperitoneoscopic versus laparoscopic adrenalectomy. Br J Surg. 2012 Dec;99(12):1639-48. doi: 10.1002/bjs.8921. Epub 2012 Sep 28. PMID 23023976
- [Background] Rubinstein M, Gill IS, Aron M, Kilciler M, Meraney AM, Finelli A, Moinzadeh A, Ukimura O, Desai MM, Kaouk J, Bravo E. Prospective, randomized comparison of transperitoneal versus retroperitoneal laparoscopic adrenalectomy. J Urol. 2005 Aug;174(2):442-5; discussion 445. doi: 10.1097/01.ju.0000165336.44836.2d. PMID 16006861
- [Derived] Barczynski M, Konturek A, Nowak W. Randomized clinical trial of posterior retroperitoneoscopic adrenalectomy versus lateral transperitoneal laparoscopic adrenalectomy with a 5-year follow-up. Ann Surg. 2014 Nov;260(5):740-7; discussion 747-8. doi: 10.1097/SLA.0000000000000982. PMID 25243546